CLINICAL TRIAL: NCT07183033
Title: Exploratory Trial on the Mechanisms of VR Intervention in Promoting Neuroplasticity Among Older Adults With Cognitive Frailty
Brief Title: Exploratory Trial of VR Intervention on Neuroplasticity in Older Adults With Cognitive Frailty
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Zheng Li, Professor, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-248
Record Dates: First submitted 2025-09-03; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Frailty
Keywords: cognitive frailty; virtual reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-Based Resistance Training Intervention (Experimental): Participants in the intervention group will receive training using a self-developed VR-based resistance training system named "Kitten Crossing the Bridge." This system primarily emphasizes static lower-limb resistance control and integrates mechanisms of task rhythm regulation, spatial judgment, and visual feedback. Preliminary usability testing has demonstrated good immersion, safety, and acceptability among older adults.The intervention will last for 4 weeks, with two sessions per week; each session will last approximately 20 minutes (excluding device setup and rest intervals). All sessions will be supervised by trained staff to ensure safety and provide necessary assistance.
  Interventions: Behavioral: VR-Based Resistance Training Intervention
- Standardized Leg-Raising Training (Active Comparator): Participants in the control group will perform standardized leg-raising exercises. The training rhythm will be guided by pre-recorded verbal prompts and demonstration videos developed by the research team, ensuring that the exercise intensity and pace are aligned with those of the intervention group.
  Interventions: Behavioral: Standardized Leg-Raising Training

INTERVENTIONS:
Behavioral: VR-Based Resistance Training Intervention — Participants in the intervention group will engage with a self-developed VR resistance training program entitled "Kitten Crossing the Bridge." This program is designed to guide older adults through static lower-limb resistance exercises, while integrating rhythm control, spatial judgment, and visual feedback. The intervention will be administered over 4 weeks, with two sessions per week; each session will last approximately 20 minutes (excluding equipment setup and rest periods). All training sessions will be supervised by qualified staff to ensure participant safety and provide necessary support.
  Arms: VR-Based Resistance Training Intervention
Behavioral: Standardized Leg-Raising Training — Participants in the control group will implement a standardized leg-raising exercise protocol, which is designed to match the intensity and rhythm of the VR-based intervention. Training will be guided by pre-recorded verbal prompts and demonstration videos developed by the research team, ensuring procedural uniformity. Each session will last approximately 20 minutes (excluding equipment setup and rest periods), with two sessions per week over a 4-week duration. All sessions will be supervised by trained staff, who will monitor participant adherence and ensure safety throughout the process.
  Arms: Standardized Leg-Raising Training

SUMMARY:
To investigate the effects of VR based intervention on neuroplasticity in older adults with cognitive frailty.

DETAILED DESCRIPTION:
This study is designed as a prospective, parallel-group, single-blind randomized controlled trial to be conducted at a senior care institution in Beijing from August to September 2025. Older adults with cognitive frailty will be randomly allocated using a computer-generated random sequence concealed in opaque sealed envelopes to either a VR-based intervention group or a control group. Allocation concealment will be maintained throughout the trial, and research staff responsible for data collection, assessment, and analysis will remain blinded to group assignments.

The intervention will comprise task-oriented VR activities specifically designed to stimulate cognitive and sensorimotor processes. Functional near-infrared spectroscopy (fNIRS) will be utilized to evaluate pre- and post-intervention neural activity, with a focus on cortical activation patterns, changes in network efficiency, and modulation of functional pathways.

This study aims to generate exploratory evidence regarding the mechanisms underlying VR-induced neuroplasticity in this population, thereby establishing a foundation for optimizing intervention parameters and targeting specific brain regions in subsequent large-scale trials.

ELIGIBILITY:
Inclusion Criteria:

* Frailty Phenotype (FP) score between 1 and 5
* Subjective Cognitive Decline Questionnaire (SCD-Q9) score ≥ 5
* Montreal Cognitive Assessment (MoCA) score between 15 and 25
* Activities of Daily Living (ADL) score ≤ 26
* Age ≥ 60 years
* Submit written informed consent prior to participating in the study

Exclusion Criteria:

* Clinical diagnosis of Alzheimer's disease, other dementias, or neuropsychiatric disorders (e.g., cerebrovascular disease, Parkinson's disease, history of traumatic brain injury, brain tumors, epilepsy)
* Current use of medications or addictive substances that may impair cognition
* Presence of musculoskeletal disorders (e.g., osteoarthritis, fractures), cardiovascular disease, or liver/kidney dysfunction that prevent safe participation in exercise
* Severe sensory or speech impairments that hinder communication
* Severe motion sickness or vestibular disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
fNIRS | Baseline, 2 Weeks, 4 Weeks
  Neural activity during the intervention tasks will be recorded using a functional near-infrared spectroscopy (fNIRS) imaging system. A 24-channel NirLight fNIRS device (Huairui Medical Technology Co., Ltd., China) will be employed, with light sources operating at wavelengths of 760-850 nm and a sampling rate of 10 Hz. The probe configuration will primarily cover the frontal, parietal, and parts of the temporal and occipital lobes.

SECONDARY OUTCOMES:
Cognitive function | Baseline, 4 Weeks
  The Chinese version of the Addenbrooke's Cognitive Examination Ⅲ (ACE-Ⅲ) is a validated neuropsychological instrument designed to assess objective cognitive function across five domains: attention, memory, verbal fluency, language, and visuospatial ability. The total score ranges from 0 to 100, with higher scores indicating better cognitive function.
  The Beijing version of Montreal Cognitive Assessment (MoCA) is a classical screening tool for mild cognitive impairment that evaluates seven cognitive domains: visuospatial and executive function, naming, attention, language, abstraction, delayed recall, and orientation. The total score ranges from 0 to 30, with higher scores indicating better cognitive performance.
  The Subjective Cognitive Decline Questionnaire (SCD-Q9) is a brief 9-item self-report questionnaire used to assess subjective cognitive symptoms in older adults. The total score ranges from 0 to 9, with higher scores reflecting more severe subjective cognitive decline.
Frailty | Baseline, 4 Weeks
  Frailty will be evaluated using the Fried phenotype model, which defines physical frailty according to five components: slowness (gait speed), weakness (hand grip strength), unintentional weight loss, exhaustion, and low physical activity. Each component is scored as present or absent, and the total score ranges from 0 to 5. A score of 0 indicates non-frail, 1-2 indicates pre-frail, and 3 or more indicates frail. Higher scores reflect more severe frailty.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No